CLINICAL TRIAL: NCT07142135
Title: Long-term Systematic Follow-up of Patients With Klinefelter Syndrome Followed at the Department of Growth and Reproduction, Rigshospitalet
Acronym: FOXXY
Status: Enrolling by invitation | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lise Aksglæde, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: H-24071762
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter syndrome; sex chromosome
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Klinefelter syndrome
  Interventions: Other: There is no intervention, only clinical description

INTERVENTIONS:
Other: There is no intervention, only clinical description — There is no intervention, only clinical description

SUMMARY:
Klinefelter syndrome (KS) is the most frequent sex chromosome disorder affecting approximately 1:660 newborn boys. The prevalence of KS rises to 3-4% among infertile males and 10-15% in patients with non-obstructive azoospermia. KS is highly underdiagnosed, and diagnosis is often delayed. Phenotypic variability, and especially a presentation with mild clinical features, often leads to diagnostic delay or non-diagnosis. It has been estimated that 50-75% of males with KS never obtain a diagnosis (Berglund et al., 2019; Bojesen et al., 2003).

Despite increasing interest in studying KS during recent years there remain significant gaps in our overall understanding of KS, including when and how to start testosterone replacement therapy (TRT), how to prevent co-morbidities, mechanisms of complications, success of fertility preservation and assessment of quality of life in affected individuals. This translates into differences in standards of care for these patients, with substantial variability in clinical practice. International guidelines regarding the care of patients with KS were published by the European Academy of Andrology/European Society of Endocrinology in 2021 (Zitzmann et al., 2021) to improve the clinical care of these patients. These guidelines, however, are limited by a general lack of scientific evidence due to the low number of studies in the field. This increases the need to systematically collect more information to develop individualized and optimized care for future patients.

The investigators therefore aim to systematically describe the phenotype of Klinefelter syndrome throughout life by collecting clinical, biochemical, genetic, and radiological data on reproductive development, fertility, anthropometry, bone age, body composition, bone mineralization, co-morbidities, biomarkers of general health as well as psychopathology and mental health.

Hypotheses:

1. Patients with KS may differ from controls in their biological health profile (hormonal, thyroid, metabolic, inflammatory, genetic, and epigenetic) which may affect their lifestyle and alter disease risk. Detailed knowledge about such alterations and at what age they appear may facilitate more individualized and optimized treatment regimens with the goal to prevent co-morbidities.
2. Hypertension, bradycardia and long QTc may be more frequently present in adults with KS. The investigators hypothesise that both blood pressure and electro cardiograph (ECG) are normal in childhood and adolescence. Knowledge about the mechanisms behind these phenomena and when they appear will help us in understanding the biological mechanism and in optimizing preventive interventions.
3. Men with KS are taller than their genetic potential. This may at least in part be attributed to an increased growth velocity through childhood before puberty.
4. Genetic and epigenetic alterations may explain the phenotypic variability and the associated co-morbidities may be caused by such alterations.
5. Virilization (penis length and width, pubic hair development, voice frequency) is impaired in adolescents and adults with KS.
6. Patients with KS face a greatly increased risk of being affected by psychopathology such as attention deficit and hyperactivity disorder (ADHD) and depression. In addition to the clinically observable lack of energy (fatigue) and social withdrawal, this may affect quality of life, and impact long-term mental health. Learning more about the factors supporting mental health in boys and men with KS will significantly advance our chances of alleviating these common complaints and preventing long-term complications.
7. Patients with KS may have distinct facial characteristics. Knowledge about such characteristics may increase the likelihood of identifying patients with KS and thereby improve the diagnostic delay.

Data Collection The data base will consist of clinical and biochemical data and results obtained at the routine control visits and admittance at a hospital. Data will be collected both retrospectively (from the medical record) and prospectively. Retrospective data from the medical record will include data collected at previous visits at the Department of Growth and Reproduction (e.g. anthropometry, Dual-Energy X-ray Absorptiometry (DXA) scans, bone age (including bone health index (BHI), hormone concentrations, karyotype, biomarkers of general health, blood pressure, pulse, semen quality, results of micro testicular sperm extraction (TESE) and testicular histology as well as medical treatment in general and other diagnoses/co-morbidity).

DETAILED DESCRIPTION:
This project is a combined retrospective (data from medical records) and prospective longitudinal study of a single centre cohort, which aims to consecutively include all patients (infants, children, adolescents and adults) with KS (47,XXY) including other rare variants of KS with more than one supernumerary X-chromosome (e.g. 48,XXXY; 48,XXYY; 49,XXXXY), mosaicism (e.g. 47,XXY/46,XY) and SRY-positive 46,XX-males (ICD: DQ980, DQ981, DQ982, DQ983, DQ984, DQ987).

Data Collection The data base will consist of clinical and biochemical data and results obtained at the routine control visits and admittance at a hospital. Data will be collected both retrospectively (from the medical record) and prospectively. Retrospective data from the medical record will include data collected at previous visits at the Department of Growth and Reproduction (e.g. anthropometry, DXA scans, bone age (including bone health index, hormone concentrations, karyotype, biomarkers of general health, blood pressure, pulse, semen quality, results of microTESE and testicular histology as well as medical treatment in general and other diagnoses/co-morbidity). All data and paraclinical parameters that will be collected prospectively are listed in the following. Some of the points are only relevant for children whereas others are only relevant for adolescents or adults as noted at each point. All points have been marked with an a or b to specify which evaluations are part of the standard care (a) and which are extra evaluations as part of the study (b).

1. Medical history (a): medical history (including karyotype, pubertal development (Tanner stages, gynecomastia, serum concentrations of reproductive hormones and growth factors), growth, DXA scans, testosterone replacement therapy (type, date, dose, effects and side-effects), family history, co-morbidities, medical treatment in general (type, date, dose), allergies, blood pressure, diet, exercise, education, and in adolescents and adults: semen quality, result of mTESE, testicular histology, alcohol consumption, smoking, drug abuse, employment/job.

2. Bone age including bone health index (a): x-ray of left hand is performed in growing boys to evaluate final height and bone health index.

3. Pubertal development and virilization:

(a) Tanner staging (pubic hair stage, gonadal stage), testicular volume by palpation, gynecomastia (b)Acne stage, voice frequency, penile length and penile width.

4. Anthropometry:

1. Height (cm) and sitting height (cm) as measured using a wall-mounted stadiometer and body weight (kg) by using an electronic scale. Target height will be calculated from biological parental heights (if available).
2. Arm span, head, thoracal, hip and waist circumferences (cm). Sitting height (cm) in adults.

   5. Clinical evaluation (a): Evaluation of tremor (yes/no), skeletal deformities (clinodactyly, pectus excavatum/carinatum, scoliosis, kyphosis, pes planus) and presence of hypermobility.

   6. Grip-strength (b): Evaluated by Digital hand dynamometer

   7. Body composition/bioimpedance (b) measured by Tanita MC780 MAS

   8. Blood samples:
   * Reproductive and adrenal hormones (a): follicle stimulating hormone (FSH), Luteinizing hormoner (LH), steroid metabolites (testosterone, dihydrotestosterone, androstendione, 17-hydroxyprogesterone, progesterone, 17-alfa-hydroxypregnenolone, estradiol, estrone, estrone sulfate, cortisol, 11-deoxycortisol, 21-deoxycortisol, 11-deoxycorticosterone, corticosterone, cortisone, aldosterone), sex hormone binding globulin (SHBG), inhibin B, anti-Müllerian hormone (AMH), insulin like factor 3 (INSL3)
   * Thyroid hormones (a): free thyroxin (T4) and thyroid stimulating hormone (TSH)
   * Thyroid antibodies (b)
   * Growth factors (b): Insulin-like growth factor-1 (IGF-1), IGF-2 and insulin-like growth factor binding protein-1 (IGFBP-1) to 6 and acid-labile subunit (ALS)
   * Bone turnover markers (a): 25-OH-vitamin D and calcium
   * Bone turnover markers (b): Phosphate, magnesium, PTH, alkaline phosphatase (liver and bone), osteocalcin, PINP (procollagen type I N-terminal propetide), CTX (carboxy terminal telopeptide of collagen type I), RANKL (receptor activator of nuclear factor kappa-B ligand), OPG (osteoprogeterin), Klotho, sclerostin and TRACP 5b (tartrate-resistant acid phosphatase 5b) in serum and urine
   * Insulin resistance (a): glucose and hemogolbin A1c (HbA1C),
   * Insulin resistance (b): Proinsulin and lipocalin-2
   * Inflammation (b): Mesoscale
   * Immune response (b): antibody titer of vaccines
   * Lipids (a): cholesterol and triglyceride
   * Lipdis (b): Free fatty acids and glycerol
   * Fat tissue (b): adiponectin and leptin
   * Haematology (a): Hematocrit and hemoglobin
   * Organ markes (a): Liver, kidney parameters and prostate specific antigen (PSA)
   * DNA purification (b) for genetic analysis (see separate section on genetics below)
   * RNA (b) (analysis of circulating small non-coding RNAs)

   Hormonal analyses and DNA purification are carried out at our own laboratories and standard biochemical analyses are performed at the hospital's central laboratory, all of which are DANAK certified.

   7. Genetic analyses A targeted approach will be used, and whole-genome or whole-exome sequencing will not be performed. A selected set of genetic polymorphisms in target genes with established or theoretic effects on metabolism, overweight, growth and infertility will be analyzed either by PCR genotyping or targeted sequencing (max. 200 selected genes). In addition, SNP-arrays that exclusively target common variants and not any rare variants will be used to determine the influence of common genetic variation on the observed associations.

   "Omfattende kortlægning af arvemassen" according to the list provided by National Ethics Committee (NVK) will not be performed. Since only commonly occurring variants are investigated, no random findings are expected.

   DNA methylation patterns will be analyzed by applying Illumina methylation arrays which do NOT reveal sequence information. The Illumina methylation array only reveal the level of methylation at common CpG sites and epigenetic analyses by sequencing will NOT be performed.

   8. Dual-energy x-ray absorptiometry scan (DXA) (a) A whole body (all) and regional (adults) DXA scan is performed to evaluate bone mineral density (BMD), total and regional body fat percentage and body lean mass. This scan is performed on an individual basis. Typically, the first time around 8-10 years if the boy can cooperate. Thereafter before starting TRT and one year after stating TRT. In adults a DXA scan is performed when the diagnosis is made and one year after starting TRT. Thereafter the patient is scanned on an individual basis depending on the results of the first scans. If the result is normal a scan will typically be performed every 5 years. If the scan shows reduced bone mineralization the patient will have another scan after 1, 2 or 3 years depending on the reduction.

   9. Blood pressure (a) The blood pressure is measured at every visit after the participants have been sitting and relaxing for at least five minutes. This will be carried out at the upper arm of the dominant side using a calibrated automatic sphygmomanometer. Blood pressure and pulse will be registered.

   10. Electrocardiography (ECG) (b) Standard ECG with 12 leads.

   11. Gonadal ultrasound (a) Ultrasound of the testicles is performed at the first visit after referral in adolescents and adults with KS.

   12. Breast ultrasound (b) Ultrasound of the breast will be performed to quantify the size of a gynecomastia, if present.

   13. Semen analysis (a) As part of the standard care of patients with KS, adolescents and adults can deliver a semen sample for analysis and if spermatozoa are present, they will have the possibility to cryopreserve the cells. The patient will be informed that most patients with KS have azoospermia and only very few cases with spermatozoa in the ejaculate have been reported. This is to prepare the patient for the most likely result.

   Sexual abstinence for 48 hours to 7 days is recommended prior to collection of a semen sample. The sample will be collected by masturbation, primarily in a designated room at the department using standard equipment.

   14. Micro TESE (a) Patients with KS older than 18 years with a fertility wish can have an operation performed (micro TESE (testicular sperm extraction)) with the goal to cryopreserve potential intratesticular spermatozoa for future fertility treatment. This is part of the standard care of patients with KS. If the patient has a history of cryptorchidism a standard testicular biopsy for histological evaluation is performed as part of the operation. This biopsy is performed to rule out the presence of precursors for testicular cancer (germ cell neoplasia in situ (GCNIS)).

   15. Questionnaires (b) A variety of questionnaires will be used to measure psychopathology and mental health in our samples. Depending on the cut-off for the individual rating scales described below, self-report forms will be used for ages 16-18 and older. For children and adolescents younger than this, parents or caregivers will respond. None of the questionnaires are diagnostic and will NOT reveal severe psychopathology that needs to be handled acutely. If concerns arise regarding issues such as poor well-being or potential signs of ADHD the family or the patient will be contacted and guided to seek appropriate help, primarily through the general practitioner who can refer for relevant follow-up care.

   To ensure valid responses in the adult self-report questionnaires assessing psychopathology and mental health, participants will be screened with a short form of the Weschler Adult Intelligence Scale, ed. 4 (WAIS-IV; (Wechsler, 2008)). On the basis of the two subtasks chosen (Vocabulary and Block Design), a mean scale score will be calculated. Mean scale scores ≥ 7 will be taken to reflect overall intellectual capacity within the normal range.

   BASC-3 Bess (Reynolds, 2015) is a 28-item rating scale designed to screen the social and psychological functioning of children and adolescents.

   ADHD-rs (DuPaul, 1998) and ASRS v.1.1 (Kessler, 2005)are brief rating scales to assess symptom characteristics of ADHD (inattention and impulsivity) in children, adolescents, and adults.

   Peds-Ql Multidimentional Fatigue Scale (Varni, 2002; Varni & Limbers, 2008) measure perceived lack of energy (fatigue) in children, adolescents, and adults.

   Brief-2 and Brief-A (Gioia, 2015) assess executive function in children, adolescents, and adults. Brief-domains address the ability to regulate emotion, attention, and behavior.

   Symptom Checklist-90 revised (SCL-90-R, (Derogatis, 1994) is a self-report inventory for adults that assesses a broad range of psychological problems and symptoms of psychopathology.

   The Autism Spectrum Quotient (Baron-Cohen et al., 2001)is a self-report questionnaire for adults designed to measure the degree to which an adult has traits associated with the autism spectrum.

   The World Health Organization Quality of Life - BREF (WHO, 1997) is a self-report questionnaire for adults which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment

   16. 3D-scan of face (b) Clinical photo including 3D-scan of face for detailed description of the facial characteristics will be performed by a LifeViz camera from QuantifiCare.

   17. Collection of biological material for a research biobank: Serum, purified DNA and urine will be stored at -20 degrees Celcius or -80 degrees Celcius after each visit. Analyses that are not part of the routine evaluation will be performed simultaneously to avoid influence of interassay variation. DNA will be purified before freezing. The research biobank consists of -20 and -80 degrees Celcius degree freezers located at Rigshospitalet in a locked room. The freezers are equipped with an alarm.

   18. Collection of biological material for a research biobank for future research: When the above-mentioned analyses have been run the exceeding material will be transferred to a biobank for future studies. The investigators aim at examining endocrinological, biochemical, metabolic, inflammatory, genetic, and epigenetic biomarkers during mini-puberty, pubertal transition as well as before and during TRT. After transferring the exceeding material to the biobank for future research the material will be stored at the Department of Growth and Reproduction for 20 years and any remaining material will be destroyed thereafter.

   The biobank can only be used for future research after new approval by the local ethics committee. When consenting to participate in the study the patient and/or family will be asked permission to save the biological material in the biobank for future studies. If the patient or the parents do not agree on saving the material in the biobank for future studies, no extra material will be saved.

   The patient or family can at any time decide that they do no longer want to have biological material stored or that they do no longer want to collect material for the biobank. In the first case all collected material will be destroyed. In the latter case no biological material will be collected in the future. Such decision will not have any consequences for the patients follow up or treatment in the department.

ELIGIBILITY:
Inclusion Criteria:

* Patients with karyotype 47,XXY or variants as mentioned above who are followed at the Department of Growth and Reproduction, Rigshospitalet, Denmark, can be included in the study.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 300 patients with these diagnoses are currently followed at The Department of Growth and Reproduction and are eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
DXA scan | DXA will be performed once
  Whole body DXA scan

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Department of Growth and Reproduction, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided